CLINICAL TRIAL: NCT04609436
Title: Clinical Use of the SmartCardia Wireless Recorder as a Telemetry System in Patients Hospitalized Outside Intensive Care (the SMART-TEL Study Trial)
Brief Title: SmartCardia Wireless Recorder as a Telemetry System
Acronym: SMARTTEL
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Stephane Cook, Professor, University Hospital Freiburg
Other Study IDs: CER 2020-0141
Record Dates: First submitted 2020-09-29; First posted 2020-10-30 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Arrhythmias, Cardiac; Monitoring
Keywords: non invasive monitoring
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: This is a single arm trial. The patient is his own control.
  Interventions: Device: Cardiac monitoring with the wireless device "SmartCardia"

INTERVENTIONS:
Device: Cardiac monitoring with the wireless device "SmartCardia" — Monitoring of arrhythmia with a wireless device (SmartCardia)

SUMMARY:
Patients hospitalized at the clinic Cecil who need telemetry will be monitored for 48 hours with the SmartCardia system in addition to conventional monitoring.

DETAILED DESCRIPTION:
Cardiac arrhythmias, such as atrial fibrillation or ventricular arrhythmias, are often asymptomatic and sometimes associated with an adverse event, such as a stroke or syncope. Telemetry monitoring in hospitals, 24 hours a day, is the most used method for detecting these cardiac arrhythmias, especially after major surgery or cardiac surgery. Currently this cardiac monitoring is ensured by a system called telemetry, a kind of box connected to 4 electrodes stuck on the patient's chest. Information is continuously transmitted to a screen located in the nurses' room, which is supposed to watch the screen continuously. There are also alarms that can be triggered when an arrhythmia occurs. In practice, it is found that very often the electrodes are disconnected for practical reasons (patient going to the toilet for example) or accidentally. The alarms are not always observed because they very often sound badly. In addition, 24-hour telemetric monitoring sometimes fails to detect the culprit arrhythmia. Event monitoring significantly increases performance of the system. It has recently been shown that the ZIO patch (iRhythm Technologies Ltd.), a wireless electrocardiography allows te detection of arrhythmias in children, confirming the usefulness of such devices in daily practice.

3.2 Investigational product and indication.

The SmartCardia patch (SmartCardia, EPFL (Ecole polytechnique fédérale Lausanne) Innovation Park, Lausanne, Switzerland) is a lightweight wireless ECG device (Figure 1) mounted on a patch with waterproof properties. The device is completely wireless and has no external connection wires. It allows patients to go about their daily activities with minimal disruption. The SmartCardia system allows in hospital patients monitoring, and corresponds to telemetry, functioning as 24 hour cardiac monitoring. The device is placed on the upper left part of the patient's chest (Figure 2). The patch can wirelessly communicate the data to a screen that will display it live. In addition, this data will be stored in the recording device and in the cloud. Once monitoring is complete, the data remains stored in the cloud and is available to physicians. During the recording, at any time, the doctor can be connected and interrogate the device in order to visualise the arrhythmias of his patient. The first studies using this device in the clinic have recently been published with very encouraging results. The device is classified in category A (Swiss government office decision attached). Previous trials with this device have shown its clinical usefulness in the intensive care unit and in daily practice. The device is actually proposed and used by many cardiologists as an alternative to the conventional Holter monitoring system. The goal of the present trial is mainly to confirm tha ability of this device to be used as a telemetry system on the ward in order to overpass the inconvenience of the actual system related to permanent cable connections with the risk of disconnexion and lost of monitoring. This trial is mainly a confirmation of that the device is a valuable option for telemetry.

The device used for this trial is the one certified by Swissmedics with UE (Union Européenne) certification

3.3 Pre-clinical evidence

The benefits of using such a type of monitoring are obvious. The patient is autonomous in his movements. The risks associated with disconnection are nonexistent. In addition, the doctor can consult the patient's data directly at any time. Finally, the data are stored in the cloud and archiving is made easier. The only risk associated with this system is an allergy to the adhesive patch. In view of the potential benefits expected from the use of this system, it is easy to understand that the study is justified. It should be kept in mind that the conventional system also has limits essentially linked to the risk of cable disconnection.

The risk linked to a bad registration of the SmartCardia system which would generate an incorrect treatment does not exist, because the clinical decision will be taken by the doctor and based only on the data provided by conventional monitoring.

Previous trials have shown the accuracy and advantages of this new wireless recorder. The system is already used in the daily practice in several countries as an alternative to conventional Holter monitoring.

3.4 Explanation for choice of comparator

The new system will be used in parallel with the conventional monitoring system. It is obvious that the conventional monitoring system should be used as the gold standard.

3.5 Risks/Benefit

There are no risks related to the use of this new device as therapeutic decision will be based only the recording of the conventional system. Benefits could be expected in the future since wireless system are preferred by the patients as demonstrated in previous trials comparing Holter monitoring and the SmartCardia device.

3.6 Justification of choice of study population

Patients after cardiac surgery are usually monitored for a few days when they are back to the ward. It is obvious that they are the cohort of choice for such monitoring since they require it anyway.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who needs to be monitored for at least 48 hours can be included in the study.

Exclusion Criteria:

* allergic to sticking plaster
* refusing to participate will be excluded from the study.
* planed MRI examination
* open wound
* Severe thorax deformity making recording not possible.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring cardiac monitoring after heart surgery will be included
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmia counting after heart surgery | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  The primary outcome is to detect supra-ventricular and ventricular arrhythmias following cardiac surgery. The following data will be reported:
  1. Number per minute of ventricular and/or supra-ventricular extrasystoles,
  2. Number per minute of supra-ventricular and/or ventricular doublets,
  3. Number per minute of supra-ventricular and/or ventricular triplets,
  4. Number of episodes/24 hours of supra-ventricular and/ot of ventricular tachycardia (VT) will be measured,
  5. Number of episodes of atrial fibrillation will be measured.
  6. Number of pause exceeding 2 seconds will be reported.

SECONDARY OUTCOMES:
Duration of arrhythmias after heart surgery | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  1. Duration of the arrhythmia will be reported in seconds.
  2. Duration of episodes of atrial fibrillation will be reported in seconds.
Noise analysis | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  Noise will also be analysed. Noise is defined as parts of the ECG signal that cannot be analysed by technicians, such as a movement artefact or muscle activity in the ECG signal. It will be measured in dividing the number of uninterpretable signals by the number of interpretable signals and reported as a percentage. This noise exists both with the SmartCardia system and with the system currently used, described as the "gold standard".
  1. The number of episodes/24 h of noise will be reported.
Incidence of noise | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  1.The number of episodes of noise will be counted.
Percentage of episodes of noise. | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  1. The percentage of noise episodes and normal detected beats will calculated in percent.

OTHER OUTCOMES:
Skin tolerance evaluation | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  Skin tolerance will be assessed for both devices, with a daily clinical evaluation by a physician. In case of intolerance a dermatologist will be consulted.
  1. Size in mm of the redness, erythema and irritation.
Skin tolerance assessment (additional measures) | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  1. CRP measurement will be perform and measured in mg/L
Skin tolerance assessment (additional measures) | 48 hours following cardiac surgery part of 10 days of hospitalization post surgery.
  2. White cells number will be measured in G/L

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Goy, MD, Principal Investigator — Hirslanden Cecil
Locations (1):
- Clinique Cecil, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No